CLINICAL TRIAL: NCT07273890
Title: Prospective, Multicenter, Controlled Study on the Impact of Real-time Feedback on Red-out
Brief Title: Real-time Feedback of Red-out Within Colonoscopy Intubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AHMU-Feedback of Red-out
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Artificial Intelligence; Colonoscopy; Real-time Feedback
Keywords: Colonoscopy; Intubation; Real-time feedback; Red-out
MeSH Terms: interventions — Intelligent Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Sham Comparator): During colonoscopy intubation, AI system is used to calculate and analyze "caecal intubation time," "red-out percentage," and the "AI-based red-out avoiding score" in real-time; however, these results are not provided as feedback to the operating colonoscopist.
  Interventions: Other: AI system
- Group B (Experimental): During colonoscopy intubation, AI system is used to calculate and analyze "caecal intubation time," "red-out percentage," and the "AI-based red-out avoiding score" in real-time, with only the caecal intubation time being provided as feedback to the operator, while the red-out percentage and AI-based red-out avoiding score are withheld.
  Interventions: Other: AI system
- Group C (Experimental): During colonoscopy intubation, AI system is used to calculate and analyze "caecal intubation time," "red-out percentage," and the "AI-based red-out avoiding score" in real-time, with only the red-out percentage being provided as feedback to the operator, while the caecal intubation time and AI-based red-out avoiding score are withheld.
  Interventions: Other: AI system
- Group D (Experimental): During colonoscopy intubation, AI system is used to calculate and analyze the "caecal intubation time" "red-out percentage," and "AI-based red-out avoiding score" in real-time, with all three results provided as feedback to the operating colonoscopist.
  Interventions: Other: AI system

INTERVENTIONS:
Other: AI system — AI-system Performance Feedback in group B, group C, and group D.

SUMMARY:
This study will employ a prospective, multicenter, controlled design. It will be conducted across multiple centers, with participated centers randomly assigned to one of four groups: Group A, Group B, Group C, and Group D.

The research will primarily focus on the AI-based analysis of colonoscopic images to calculate the following metrics: caecal intubation time, red-out percentage, and the AI-based red-out avoiding score. Based on the study's implementation protocol, a decision will be made regarding whether to provide real-time feedback. Additionally, the presence of any complications will be assessed both during and after the colonoscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Study Participants (Patients):

   Aged 18 to 70 years, any gender. Individuals scheduled to undergo diagnostic or screening colonoscopy at the investigational site.
2. Colonoscopists:

Expert-level colonoscopists (having performed a total of >1000 colonoscopy procedures).

Right-handed.

Exclusion Criteria:

1. Study Participants (Patients):

   Individuals undergoing the following procedures:

   cases with a history of colorectal surgery; cases with a history of chemotherapy, raditherapy; cases with a history of abdominal, and/or pelvic surgery; cases with a history of difficult colonoscopies; cases with colorectal tumours and obstructive lesions; cases with colorectal diverticula; cases with ulcerative colitis or Crohn's disease; cases with ischemic bowel disease; cases with colorectal polyposis; cases with melanosis coli; cases undergoing sigmoidoscopy; cases with poor intestional cleanliness (segment Boston bowel preparation scale (BBPS) of < 2 points, total BBPS of < 6 points); cases undergoing therapy procedures such as biopsy or CSP during the intubation phase; cases with transparent cap assisted colonoscopy; cases with water-assisted colonoscopy; cases with air insufflation level of M or L; cases failed caecal intubation within 15 min; cases with colonoscope stiffness level > 0; obese cases or underweight cases; and cases refusing participation.

   Individuals who decline to provide informed consent.
2. Colonoscopists:

Those who have performed fewer than 300 complete colonoscopies in any calendar year within the past three years.

Those who decline to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-04-20 (Estimated)

PRIMARY OUTCOMES:
Red-out percentage | Stage 3 (projected to begin in 3-6 months)
  The impact of real-time feedback on red-out percentage.
Caecal intubation time | Stage 3 (projected to begin in 3-6 months)
  The impact of real-time feedback on caecal intubation time.
AI-based red-out avoiding score | Stage 3 (projected to begin in 3-6 months)
  The impact of real-time feedback on AI-based red-out avoiding score.

SECONDARY OUTCOMES:
Complications | Stage 3 (projected to begin in 3-6 months)
  During and after the colonoscopy, assess for any signs of complications